CLINICAL TRIAL: NCT01415141
Title: A Randomized Trial of Telaprevir, Peginterferon, and Ribavirin Versus Peginterferon and Ribavirin for Treatment of Genotype 1 Hepatitis C Virus With Host Interleukin 28B CC Polymorphism
Brief Title: Peginterferon and Ribavirin, With or Without Telaprevir, for Genotype 1 Hepatitis C and IL28B CC Polymorphism
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Steven Lidofsky, Principle Investigator, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M11-219
Record Dates: First submitted 2011-08-01; First posted 2011-08-11 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis C
Keywords: genotype 1; IL28B CC polymorphism; telaprevir; peginterferon; ribavirin
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin; telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PR (Active Comparator): Treatment with Peginterferon and Ribavirin for up to 48 weeks
  Those who achieve eRVR will receive 24 weeks of treatment
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- TPR (Active Comparator): Treatment with Telaprevir, Peginterferon and Ribavirin. Patients will receive all 3 drugs for 12 weeks then switch to Peginterferon and Ribavirin for 36 weeks
  Those who achieve eRVR will receive 12 weeks of treatment with all 3 drugs and then 12 weeks of treatment with the 2 drugs.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin; Drug: telaprevir

INTERVENTIONS:
Drug: Peginterferon alfa-2a — 180ug subcutaneously, weekly
Drug: Ribavirin — Administered orally twice a day as follows:
  weight < 75kg - 1000mg weight ≥ 75kg - 1200mg
Drug: telaprevir — 750mg every 8 hours, orally
  Arms: TPR

SUMMARY:
Chronic hepatitis C is a major cause of liver disease and is thus an important public health problem. Although some strains (genotypes) of the hepatitis C virus are highly responsive to treatment with a combination of peginterferon and ribavirin, the most common form of the virus (genotype 1) is relatively resistant to this treatment. Recently, telaprevir has been approved by the Food and Drug Administration to be given in combination with peginterferon and ribavirin. This 3-drug combination boosts the remission rate for genotype 1 hepatitis C to that seen with other more responsive hepatitis C genotypes treated with only peginterferon and ribavirin. However, telaprevir has additional side affects such as rash and anemia that may limit its usefulness. Intriguingly, about one third of patients infected with genotype 1 hepatitis C, who have a specific variation (polymorphism) in the DNA sequence (CC) near an immune response gene (IL28B), in fact are highly responsive to 2-drug treatment with peginterferon and ribavirin. This raises the possibility that individuals who have the IL28B CC polymorphism may not need to be treated with the addition of telaprevir and could therefore be spared unnecessary side effects. Thus, the purpose of this study is to determine among genotype 1 hepatitis C patients with the IL28B CC polymorphism the success rate and side effects of 3-drug treatment compared with 2-drug treatment.

In this study, patients with genotype 1 chronic hepatitis C who have the IL28B CC polymorphism will be randomly assigned to be treated with telaprevir, peginterferon, and ribavirin or with only peginterferon with ribavirin. These medications and the procedures involved, including patient history, physical examination, and obtaining small volume blood specimens (less than 4 teaspoons) for laboratory testing, are within the scope of standard management of hepatitis C treatment. All patients will be monitored during treatment with periodic blood testing (weeks 2, 4, and every 4 weeks thereafter while on treatment, and 24 weeks after stopping treatment) and office visits (weeks 5, 12, 25, 49 while on treatment and 25 weeks after stopping treatment). The success of treatment will be judged by the presence or absence of detectable virus in blood, as measured by a sensitive diagnostic test (PCR). The data to be generated will include measurement by PCR of hepatitis C viral loads before, during, and after treatment, as well as reporting of adverse drug effects.

DETAILED DESCRIPTION:
Chronic infection with the hepatitis C virus (HCV), which affects 1-2% of adults in the United States, is a major risk factor for liver failure due to cirrhosis and/or hepatocellular carcinoma (Davis 2010). Epidemiological information suggests that the frequency of these HCV-related sequelae is likely to continue to increase over the next 10-15 years unless effective and well-tolerated treatments become available. Development of improved antiviral therapy is thus an important public health priority.

Until recently, the most effective treatment for chronic HCV infection has been a combination of peginterferon and ribavirin, given for up to 48 weeks. With this regimen, the sustained virological response (SVR), defined as undetectable HCV RNA 24 weeks after completion of antiviral treatment, is approximately 50-60% (Hoofnagle 2006). Not all patients are able to complete therapy however; up to 10% will discontinue this prematurely as a result of intolerable side effects, predominantly depression and/or fatigue (Seeff 2010). The major determinants of responsiveness to antiviral therapy are viral genotype and selected host characteristics. Hepatitis C genotype 1 (HCV-1), which accounts for approximately 70% of chronic infections in North America, and is relatively resistant to treatment with peginterferon and ribavirin. SVR with treatment for HCV-1 is approximately 40% (Hoofnagle 2006). That said, among HCV-1-infected individuals, there is diversity in SVR, which is correlated with a dinucleotide polymorphism at a locus upstream of the interleukin 28B (IL28B) gene. Specifically, with 48 weeks of peginterferon and ribavirin therapy, 70% of individuals with the IL28B CC polymorphism achieve SVR, compared with only 30% of individuals with other IL28B polymorphisms (Thompson 2010).

New treatments for chronic HCV-1 infection are now available. In May 2011, the Food and Drug Administration (FDA) approved telaprevir, an orally available small molecule inhibitor of the HCV-1 protease, for treatment of chronic HCV-1, to be given in combination with peginterferon and ribavirin. In HCV-1-infected patients, this three-drug regimen has been shown to confer an SVR of 75% (Jacobson 2011). However, this regimen appears to be associated with up to a nearly 1.5-fold increase in premature drug discontinuation, in comparison with a regimen of peginterferon, and ribavirin alone, largely influenced by the development of telaprevir-associated rash. Given the high responsiveness to conventional peginterferon and ribavirin among HCV-1-infected individuals with the IL28B CC polymorphism, we hypothesize SVR will not be enhanced in such individuals by the addition of telaprevir to peginterferon and ribavirin therapy. If this is correct, HCV-1-infected patients with the IL28B CC polymorphism can then be treated with comparable success with peginterferon and ribavirin alone and will therefore be spared telaprevir-associated adverse affects.

The proposed study, which is a prospective randomized open label trial (in HCV-1-infected subjects with the IL28B CC polymorphism) of treatment with telaprevir (T), peginterferon (P), and ribavirin (R) versus PR alone, will test the working hypothesis. The study design takes advantage of the concept of response-guided treatment, a strategy in which the duration of antiviral treatment is based upon the presence or absence of a rapid virological response (RVR), defined as loss of detectable serum HCV RNA within the first 4 weeks of therapy. In particular, it has been shown that HCV-1 patients who achieve RVR (and maintain undetectable HCV RNA at 12 weeks (defined as eRVR), with either PR-containing or TPR-containing regimens have comparable SVR with 24 weeks, compared with 48 weeks, of total treatment (Mangia 2008, Jacobson 2011).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Serum Hepatitis C RNA > 10,000IU/mL
* Hepatitis C virus genotype 1
* IL28B polymorphism

Exclusion Criteria:

* Previous treatment for chronic Hepatitis C
* clinical or biological evidence of acute hepatitis, including serum ALT or AST > 300U/ml
* HIV antibody positive, hepatitis b surface antigen positive or known diagnosis of other chronic liver disease
* Contraindications to PR-based treatment:

  1. uncontrolled psychiatric illness
  2. active substance dependency
  3. Known autoimmune disorder
  4. Untreated thyroid disease
  5. Uncontrolled seizure disorder
  6. Pregnancy, lactation or inability to maintain contraception
  7. Chronic kidney disease w/ estimated GFR< 60
  8. ANC<1.5/nl, Hb<12g/dl, or platelets<75/nl
* Clinical or biochemical evidence of decompensated liver disease including:

  1. History of encephalopathy, ascites, or variceal bleeding OR
  2. Bilirubin > 3g/dl or INR > 1.5
* Life threatening disorder with expected median survival less than 5 years
* Inability to comply with drug regimens or testing schedule required for study
* Lack of insurance coverage for any of the study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Sustained virological response among subjects receiving a three drug versus two drug regimen of treatment | 24 weeks after completion of treatment
  Sustained virological response is defined as undetectable hepatitis C virus RNA in the blood at 24 weeks after the completion of antiviral treatment. This will be measured by PCR to determine the hepatitis C viral load in blood at the indicated time point.

SECONDARY OUTCOMES:
Extended rapid virological response in patients receiving three drug versus two drug regimen | weeks 4 and 12 of treatment
  Extended rapid virological response (eRVR) is defined as undetectable hepatitis C virus RNA in the blood at 4 and 12 weeks of treatment. This will be measured by PCR to measure viral load at the indicated time points.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lidofsky, MD, Principal Investigator — University of Vermont & Fletcher Allen Health Care
Locations (2):
- United States (2):
  - Emory University School of Medicine, Atlanta, Georgia
  - Fletcher Allen Health Care, Burlington, Vermont

REFERENCES:
- [Background] Davis GL, Alter MJ, El-Serag H, Poynard T, Jennings LW. Aging of hepatitis C virus (HCV)-infected persons in the United States: a multiple cohort model of HCV prevalence and disease progression. Gastroenterology. 2010 Feb;138(2):513-21, 521.e1-6. doi: 10.1053/j.gastro.2009.09.067. Epub 2009 Oct 25. PMID 19861128
- [Background] Hoofnagle JH, Seeff LB. Peginterferon and ribavirin for chronic hepatitis C. N Engl J Med. 2006 Dec 7;355(23):2444-51. doi: 10.1056/NEJMct061675. No abstract available. PMID 17151366
- [Background] Mangia A, Minerva N, Bacca D, Cozzolongo R, Ricci GL, Carretta V, Vinelli F, Scotto G, Montalto G, Romano M, Cristofaro G, Mottola L, Spirito F, Andriulli A. Individualized treatment duration for hepatitis C genotype 1 patients: A randomized controlled trial. Hepatology. 2008 Jan;47(1):43-50. doi: 10.1002/hep.22061. PMID 18069698
- [Background] Seeff LB, Ghany MG. Management of untreated and nonresponder patients with chronic hepatitis C. Semin Liver Dis. 2010 Nov;30(4):348-60. doi: 10.1055/s-0030-1267536. Epub 2010 Oct 19. PMID 20960375
- [Background] Thompson AJ, Muir AJ, Sulkowski MS, Ge D, Fellay J, Shianna KV, Urban T, Afdhal NH, Jacobson IM, Esteban R, Poordad F, Lawitz EJ, McCone J, Shiffman ML, Galler GW, Lee WM, Reindollar R, King JW, Kwo PY, Ghalib RH, Freilich B, Nyberg LM, Zeuzem S, Poynard T, Vock DM, Pieper KS, Patel K, Tillmann HL, Noviello S, Koury K, Pedicone LD, Brass CA, Albrecht JK, Goldstein DB, McHutchison JG. Interleukin-28B polymorphism improves viral kinetics and is the strongest pretreatment predictor of sustained virologic response in genotype 1 hepatitis C virus. Gastroenterology. 2010 Jul;139(1):120-9.e18. doi: 10.1053/j.gastro.2010.04.013. Epub 2010 Apr 24. PMID 20399780
- [Background] Jacobson IM, McHutchison JG, Dusheiko G, Di Bisceglie AM, Reddy KR, Bzowej NH, Marcellin P, Muir AJ, Ferenci P, Flisiak R, George J, Rizzetto M, Shouval D, Sola R, Terg RA, Yoshida EM, Adda N, Bengtsson L, Sankoh AJ, Kieffer TL, George S, Kauffman RS, Zeuzem S; ADVANCE Study Team. Telaprevir for previously untreated chronic hepatitis C virus infection. N Engl J Med. 2011 Jun 23;364(25):2405-16. doi: 10.1056/NEJMoa1012912. PMID 21696307